CLINICAL TRIAL: NCT04055974
Title: Promoting Maternal Mental Health: Applicability and Effectiveness of an eHealth Intervention for Portuguese Postpartum Women
Brief Title: Be a Mom: Effectiveness of an eHealth Intervention for Promoting Maternal Mental Health
Acronym: BeAMom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Ana Fonseca, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SFRH/BD/115585/2016
Record Dates: First submitted 2019-07-23; First posted 2019-08-14 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Mental Health Wellness 1
Keywords: positive mental health; cognitive behavioral therapy; eHealth; postpartum period

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single-blind - the investigator is unaware of the intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BeAMom (Experimental): Low-risk (LR) women will receive a web-based intervention for the promotion of maternal mental health (the Be a Mom program). In addition, women will receive postpartum treatment as usually performed in primary care settings (TAU).
  Interventions: Behavioral: Be a Mom
- Control (No Intervention): Low-risk (LR) women will receive postpartum treatment as usually performed in primary care settings (TAU). During medical appointments, health professionals may ask women and provide information about psychological problems during the postpartum period.

INTERVENTIONS:
Behavioral: Be a Mom — The Be a Mom program is a web-based self-guided cognitive-behavioral intervention targeting postpartum women. It consists of 5 weekly modules, each targeting a specific thematic content, and providing women with both information and specific therapeutic strategies (with a strong focus on cognitive-behavioral techniques) to address each thematic content. Modules are sequential.
  Arms: BeAMom

SUMMARY:
Be a mom (a web-based cognitive-behavioral intervention) is being tested in another trial as a preventive intervention in the postpartum period (NCT03024645). However, given its content and the focus on developing and strengthening psychological resources, it is important to understand if Be a Mom is also effective in promoting maternal mental health of postpartum women who are not at risk of developing postpartum depression. Thus, the main goal of this research is to apply and evaluate Be a Mom for the promotion of mental health, in terms of its efficacy, acceptability and feasibility (user's adherence, dropout), user's satisfaction and cost-effectiveness.

The RCT will be a two-arm trial. Women with a child aged up to 3 months old will be enrolled in the study. A minimum number of 1000 women will be enrolled in the study. After agreeing to participate in the study, the women will be screened for the absence of risk factors for PPD (PDPI-R < 5.5). In case of a negative screen, women will be randomly assigned to one of two conditions: the intervention (Be a Mom program) or the control condition. The sample will be recruited online.

Participation in this study will last 15 months. The Be a Mom program will last 5 weeks. Participants in both conditions will be invited via email to complete baseline, post-intervention and follow-up assessments (4-months and 12-months after post-intervention). Assessments will include self-report questionnaires to assess several indicators (e.g., positive mental health, quality of life, marital satisfaction, depressive and anxiety symptoms, maternal self-efficacy), mechanisms that may be involved in the treatment response (e.g., self-compassion, emotional regulation), user's acceptability and satisfaction and cost-effectiveness.

DETAILED DESCRIPTION:
In the present study, a web-based intervention to promote women's mental health in the transition to motherhood (the Be a Mom program) will be tested. The design and content development of the Be a Mom program was conducted through a formative evaluation process.

The transition to motherhood is a widely studied period that is characterized as demanding for mothers, and that entails an adjustment to lifestyle changes and new responsibilities. There is extensive research suggesting that this period is a time of increased risk for psychological problems, such as postpartum depression. In turn, this can lead to numerous negative consequences to the mother and the child's development.

Even women who are not at an immediate risk of developing postpartum depression face numerous challenges and concerns that may place them in a vulnerable position (e.g., health needs, infant care, conflict with partner, changes in marital/social relationships, transitioning back to work). Despite this, research on the transition to motherhood has largely focused on women at risk or presenting mental illness, overlooking all women in the postpartum period and their positive mental health.

Evidence shows that positive mental health over time functions as a resilience resource and protects against both physical and mental illness. There is also evidence suggesting that the lack of positive mental health may also make individuals more vulnerable to future adversities. This implies that the promotion of positive mental health should be an additional goal in public and mental health care that complements the treatment of psychopathology.

Be a Mom is self-guided web-based intervention grounded on CBT principles that also includes recent developments in acceptance and commitment based-therapies, specifically for the perinatal context. This program focuses on the development and enhancement of psychological resources such as self-compassion and psychological flexibility and an increase of mental health literacy. Be a Mom has a modular set-up that is updated weekly, with each module addressing one or two specific thematic contents (Changes and reorganizations during the transition to parenthood; Emotional diversity; Cognitions; Relationship with others [social support and communication]; Couple relationship; Signs and symptoms of depression and help-seeking). In each module, participants will be provided with both psychoeducational content and therapeutic strategies. Informational material will be given in text format, combined with audio, video and/or animations. The Be a Mom program will also include interactive tools and feedback tools to support learning.

The main goal of the research is to apply and evaluate Be a Mom for the promotion of maternal mental health, in terms of its efficacy, acceptability and feasibility (user's adherence, dropout), user's satisfaction and cost-effectiveness. The efficacy of the program will be assessed considering two indicators: a) increase in levels of positive mental health at post-intervention and throughout the first postpartum year; and b) post-intervention and follow-up improvements in mother's psychosocial adjustment indicators (e.g., depressive and anxiety symptoms, self-empowerment, quality of life, maternal self-efficacy, marital satisfaction). The present study will also aim to investigate the mechanisms explaining the treatment response (e.g., self-compassion, emotion regulation).

The research design of the trial followed the methodological recommendations for the development and evaluation of web-based interventions. A pilot study was conducted in order to assess user's satisfaction and acceptability of the structure and content of the Be a Mom program and carry out appropriate adjustments. The results allowed to identify and implement modifications and the final version of Be a Mom was conducted, allowing for further efficacy studies.

The RCT will be a two-arm prevention trial, conducted in low-risk women (PDPI-R < 5.5). The intervention condition (the Be a Mom program) will be compared with a control condition (Treatment as Usual). The sample will include women who delivered a healthy baby in the early postpartum period (up to 3 months postpartum). Women will be recruited online through social media and websites and forums focused on motherhood. A minimum number of 150 women per condition will be required (N=300). Accounting for the proportion of high-risk and low-risk women and the 50% of attrition rate over time, an anticipated sample of 1000 women will be enrolled in the study.

Women who demonstrate interest in the study will be informed of the study goals, the structure and arms of the research and the researchers' and participants' roles. Women who agree to participate in the study will give their informed consent. All ethical requirements for research with humans are guaranteed. Women will be screened for the presence of risk factors for PPD. In case of presence of risk factors, women's participation in the study will end. In case of not presenting risk factors for PPD (PDPI-R < 5.5), women be randomly assigned (blocked randomization, with allocation concealment) to one of the conditions: the intervention (Be a Mom program) or the control condition.

A researcher (licensed psychologist) will contact women in the intervention condition, aiming to explain the program's structure and provide assistance during the course of the study.

Participation in the study will last 15 months. The Be a Mom program will last 5 weeks. Participants in both conditions will be invited via email to complete baseline, post-intervention and follow-up (4-months and 12-months after post-intervention) assessments. Assessments will include self-report questionnaires to assess several indicators (e.g., mental health, quality of life, marital satisfaction, depressive and anxiety symptoms, maternal self-efficacy), mechanisms that may be involved in the treatment response (e.g., self-compassion, emotional regulation), user's acceptability and satisfaction and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Having 18 years or more;
* Being female;
* Having had a live healthy birth in the last 3 months, with both woman and the child discharged from hospital;
* Internet access at home.
* Absence of risk factors for Postpartum Depression (PDPI-R < 5.5).

Exclusion Criteria:

* Current diagnosis of serious mental health condition (e.g., substance abuse, bipolar disorder);
* Currently receiving treatment for depressive symptoms, including antidepressant medication or psychotherapy;
* Language difficulties that impede comprehension/reading-writing;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in the presence of positive mental health | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with Mental Health Continuum-SF (MHC-SF; Keyes et al., 2008). The MHC-SF can be scored continuously (scores range from 0 to 70, and higher scores indicate better positive mental health) or categorically considering mental health status (flourishing, moderate mental health, languishing)

SECONDARY OUTCOMES:
Changes from baseline in depressive symptoms | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with Edinburgh Postnatal Depression Scale (EPDS; Cox et al., 1997). The total score ranges between 0 and 30, and higher scores are indicative of more severe depressive symptoms.
Changes from baseline in anxiety symptoms | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with the Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS; Snaith & Zigmond, 1994). The total score ranges between 1 and 28, and higher scores are indicative of more severe anxiety symptoms.
Changes from baseline in self-empowerment | From baseline to postintervention (8 weeks after randomization); 4 months postintervention
  Measured with the Self-Empowerment Scale (SES; Rogers et al., 1997). The total score ranges between 0 and 100, and higher scores are indicative of higher self-empowerment.
Changes from baseline in marital satisfaction: Marital Satisfaction Subscale of the Investment Model Scale | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with the Marital Satisfaction Subscale of the Investment Model Scale (IMS; Rusbult et al., 1998). The total score ranges between 0 and 60, and higher scores are indicative of higher relationship satisfaction.
Changes from baseline in maternal self-efficacy | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with the Perceived Maternal Parenting Self-Efficacy Questionnaire (PMP S-E; Barnes & Macedo, 2007). The total score ranges between 1 and 80, and higher scores are indicative of a higher perceived maternal self-efficacy.
Changes from baseline in psychological flexibility | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with the Acceptance and Action Questionnaire-II (AAQ-II; Bond et al., 2011). The total score ranges between 1 and 49, and higher scores are indicative of a higher psychological flexibility.
Changes from baseline in self-compassion | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with the Self-Compassion Scale-SF (SCS-SF; Raes et al., 2011). The total score ranges between 1 and 48, and higher scores are indicative of higher self-compassion.
Changes from baseline in emotional regulation | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with the Difficulties in Emotional Regulation Scale (DERS-SF; Kaufman et al., 2015). The total score ranges between 1 and 90, and higher scores are indicative of more difficulties in emotion regulation.
Parental psychological flexibility | Measured at follow-up (4 and 8 months postintervention)
  Measured with the Parental Acceptance Questionnaire (6PAQ; Greene et al., 2015). The total score ranges between 1 and 72, and lower scores are indicative of higher parental psychological flexibility.
Acceptability of the program for postpartum women: Measured through specific questions | Measured at post-intervention (8 weeks after randomization)
  Measured through specific questions (to be developed by the researchers) to assess acceptability.
Feasibility of the program for postpartum women (Measured through the website utilization) | Measured at post-intervention (8 weeks after randomization)
  Measured through the website utilization (e.g., number of logins, average visit length, total time spent on the website, number of exercises completed) and dropout rate.
Medical Costs | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with the Treatment Inventory of Costs in Psychiatric Patients (TiC-P; Hakkaart-van, 2002)
Health state and EQ-VAS | From baseline to postintervention (8 weeks after randomization); 4 and 8 months postintervention
  Measured with the Euroqol Five Dimension Scale (EQ-5D; Euroqol Group, 1990). The EQ-5D consists of 2 pages: the EQ-5D descriptive system (used to generate a health state profile) and the EQ visual analogue scale (EQ VAS - used as a quantitative measure of health outcome that reflects the patient's own judgement). Each health state can be assigned a summary index score based on societal preference weights for the health state. These weights (or utilities) are used to compute QALYS. Health state index scores range from less than 0 (0 is a health state equivalent to death, negative values are valued as worse than death) to 1 (perfect health), with higher scores indicating higher health utility. Regarding the VAS, participant rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Fonseca, PhD, Principal Investigator — University of Coimbra
Locations (1):
- Faculty of Psychology and Education Sciences, University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monteiro F, Pereira M, Canavarro MC, Fonseca A. Be a Mom, a Web-Based Intervention to Promote Positive Mental Health Among Postpartum Women With Low Risk for Postpartum Depression: Exploring Psychological Mechanisms of Change. Front Psychiatry. 2021 Jul 14;12:701107. doi: 10.3389/fpsyt.2021.701107. eCollection 2021. PMID 34335336